CLINICAL TRIAL: NCT04792593
Title: Senl-h19 CAR-T Cell Injection in the Treatment of Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Senl-h19 CAR-T for B-ALL
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: B-ALL
Keywords: B-ALL，h19，CAR-T

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senl-h19 CAR-T (Experimental): Patients will be treated with Senl-h19 CAR-T cells
  Interventions: Biological: Senl-h19 CAR-T

INTERVENTIONS:
Biological: Senl-h19 CAR-T — Biological: Senl-h19 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis
  Other Names: CD19 CAR-T

SUMMARY:
This study is an open, dose-escalating clinical study, taking patients with relapsed or refractory acute lymphoblastic leukemia as the test subjects, including mouse-derived CAR-T treatment failure or relapse, or for any reason cannot bridge the transplant r/r B-ALL.

DETAILED DESCRIPTION:
Main research objectives:

To evaluate the safety and efficacy of Senl-h19 CAR-T in patients with relapsed or refractory acute lymphoblastic leukemia Secondary research purpose To investigate the cytokinetic characteristics of Senl-h19 CAR-T in patients with relapsed or refractory acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the informed consent and be willing and able to comply with the visit, treatment protocol, laboratory examination, and other requirements of the study as specified in the study procedure sheet; 2. A definite diagnosis of relapsed and refractory acute B-lymphoblastic leukemia meets one of the following criteria: a) Mouse CAR-T treatment fails or relapses; B) Unable to bridge the graft for any reason; 3. Eastern Cooperative Oncology Group (ECOG) score ≤2; 4. Age ≥2 years old, male or female 5. CD19 positive tumor cells were detected by immunohistochemistry or flow cytometry; 6. Expected survival longer than 3 months; 7. The collection time of peripheral blood mononuclear immune cells must be at least 2 weeks from the last radiotherapy or systematic treatment of patients;

Exclusion Criteria:

* 1. Severe cardiac insufficiency; 2. Have a history of severe lung impairment; 3. Complicated with other advanced malignant tumors; 4. Complicated with severe or persistent infection that cannot be effectively controlled; 5. Complicated with severe autoimmune diseases or congenital immune deficiency; 6. Active hepatitis (HBVDNA or HCVRNA positive); Human immunodeficiency virus (HIV) infection or syphilis infection; 8. Have a history of severe allergy to biological products (including antibiotics); 9. The female patient is pregnant and lactating, or has a pregnancy plan within 12 months; 10. Conditions that the investigator believes may increase the risk to the subject or interfere with the outcome of the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD7 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

SECONDARY OUTCOMES:
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of Senl h19 CAR- T cells in the genomes of PBMC by qPCR method
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua MD Lu, PhD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei yanda Ludaopei Hospital, Yanda, Hebei, China